CLINICAL TRIAL: NCT02363101
Title: Health Outcomes and Costs (HOC) in Brazilian Public Health Care System - The HOC Study in Lung Cancer
Brief Title: Health Outcomes and Costs (HOC) in Lung Cancer (LC)
Acronym: HOC-LC
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Instituto Nacional de Cancer, Brazil (Other Government)
Collaborators: Instituto Nacional de Cardiologia de Laranjeiras (Other)
Responsible Party: Principal Investigator, Carlos Gil Moreira Ferreira, MD PHD, Instituto Nacional de Cancer, Brazil
Other Study IDs: INCA012015
Record Dates: First submitted 2015-02-09; First posted 2015-02-13 (Estimated); Last update posted 2015-03-04 (Estimated); Status verified 2015-03

CONDITIONS: Lung Cancer
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to evaluate the costs, health-related quality of life and preference values from lung cancer patients assisted in a Brazilian public health care unit.

DETAILED DESCRIPTION:
The costs will be assessed by micro-costing approach. All procedures involved in lung cancer at diagnosis, staging, treatment and best supportive care will be assessed.

The health-related quality of life will be assessed by EORTC-QLQ-C30, EQ-5D and EORTC-QLQ-LC13 in all different stages of lung cancer.

An utility measure will be considered. The preference values will be assessed via discrete choice experiment. Two scenarios will be designed and the lung cancer patients will be asked about the preferences.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of lung cancer disease
* Able to understand the overall concept of study and sign the written informed consent

Exclusion Criteria:

* Illiterate
* Visible cognitive impaired
* Non-primary lung tumor

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Lung cancer patients from Instituto Nacional de Câncer during one year.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2015-03; Primary Completion 2016-03 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Direct costs | one year
  Direct costs related to each procedure involved on lung cancer
HRQoL | up to 30 days after the procedure
Preference values | cross sectional
  Evaluate preference values in hypothetic scenarios

CONTACTS AND LOCATIONS:
Overall Officials: Carlos Gil Ferreira, Principal Investigator — National Cancer Institute, France; Luciene Schluckebier, Study Director — National Cancer Institute, France; Marisa Santos, Study Chair — INC; Bruna Carvalho, Study Chair — National Cancer Institute, France; Pedro Masson, Study Chair — National Cancer Institute, France; Andréa Monteiro, Study Chair — INC; Bruna Medeiros, Study Chair — INC; Kátia Senna, Study Chair — INC; Márcia Gisele, Study Chair — INC
Locations (1):
- INCA - Instituto Nacional de Câncer, Rio de Janeiro, Rio de Janeiro, Brazil